CLINICAL TRIAL: NCT06983912
Title: The Effect of Preoperative Rehabilitation on Functional Recovery After Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Preoperative Rehabilitation Training and Total Knee Arthroplasty Outcomes
Acronym: PRTKAO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fuzhou University Affiliated Provincial Hospital (Other)
Responsible Party: Principal Investigator, Haiqi Ding, Clinical Professor, Fuzhou University Affiliated Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: FuzhouAffiliated
Record Dates: First submitted 2025-04-26; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-04

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (No Intervention)
- Preoperative Rehabilitation Training (Experimental)
  Interventions: Behavioral: Preoperative Rehabilitation Training

INTERVENTIONS:
Behavioral: Preoperative Rehabilitation Training — Initiate preoperative Physical Rehabilitation Training (PRT) starting from the preoperative period, with training five days a week up until the day before surgery. This includes:
  Muscle Strength Training: Isometric contractions of the quadriceps, straight leg raises, etc., for 15-20 minutes per session, twice daily.
  Joint Mobility Training: Flexion and extension exercises of the knee joint, ankle pump exercises, etc., for 10-15 minutes per session, twice daily.
  Balance Training: One-legged standing, center of gravity shifting exercises, etc., for 10-15 minutes per session, twice daily.
  Activities of Daily Living Training: Transfer training from sitting to standing, walking exercises, etc., for 10-15 minutes per session, twice daily.
  Arms: Preoperative Rehabilitation Training

SUMMARY:
Joint replacement surgery is an effective treatment for severe joint diseases, but the postoperative recovery process is complex and lengthy. Preoperative rehabilitation training, as an important part of preoperative preparation, has been proven to significantly improve postoperative recovery outcomes. However, there is currently a lack of systematic research on the optimal protocols and duration of preoperative rehabilitation training and their specific impacts on postoperative recovery. This study aims to evaluate the effects of preoperative rehabilitation training on postoperative recovery after joint replacement through a randomized controlled trial, providing scientific evidence for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis is osteoarthritis and Scheduled for joint replacement surgery.
2. Age ≥18 years old and ≤90 years old, with no gender restrictions.
3. Patients voluntarily participate in the study and sign the informed consent form.

Exclusion Criteria:

1. Severe cardiopulmonary insufficiency, unable to tolerate rehabilitation training.
2. Neurological disorders leading to motor dysfunction.
3. Mental illnesses that prevent cooperation with rehabilitation training.
4. Severe joint deformities or muscle atrophy present before surgery, affecting the implementation of rehabilitation training.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Knee Joint Function Assessment | Following total knee arthroplasty, assessments are typically conducted at the 1st, 3rd, 6th, and 12th month post-surgery
  Knee injury and Osteoarthritis Outcome Score (KOSS): KOOS is a scale used to assess symptoms and function in patients with knee injury and osteoarthritis, widely applied in clinical practice and research. It includes five dimensions (pain, other symptoms, function in daily living, function in sport and recreation, quality of life), with each dimension comprising several questions that patients rate based on their personal conditions. The scoring range for each question is 0-10 points, where 0 indicates no symptoms or difficulty, and 10 indicates the most severe symptoms or difficulties. The total score for each dimension is the average of all the questions within that dimension, ranging from 0 to 100 points. The higher the score, the milder the symptoms and the better the function.

SECONDARY OUTCOMES:
Postoperative Assessment | Following total knee arthroplasty, assessments are typically conducted at the 1st, 3rd, 6th, and 12th month post-surgery.
  Aggregated Locomotor Function: ALF score is a scale designed to assess knee joint function, primarily by measuring the time it takes for patients to complete specific physical tasks to evaluate their motor function. This scale includes the following three parts: 8-meter walking time, time to climb up and down stairs, and chair transfer time. The total ALF score is obtained by adding the average time of the above three tasks. The shorter the time, the lower the score, indicating better motor function.

IPD SHARING:
Plan to Share IPD: Undecided